CLINICAL TRIAL: NCT03734523
Title: Clinical Trial to Survey Results of Flourish Vaginal Care System for Recurrent Bacterial Vaginosis
Status: Completed | Type: Observational
Sponsor: Vaginal Biome Science (Other)
Collaborators: Concord Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SAIRB-16-0013
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Bacterial Vaginosis; Vaginal Flora Imbalance
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pilot Group: 12 week study: Premenopausal women between 18 and 52 who have been diagnosed with BV at least once within the past year will be invited to enroll. They will be followed longitudinally for 12 weeks. As this is an observational study, there is no control group.
  Exclusions: pregnant women, those with allergies/sensitivities to product ingredients or to Diflucan or metronidazole, anyone who is immunocompromised, anyone with known vaginal infection other than BV or yeast, those who may be mentally/emotionally triggered by VSQ questions. We will exclude vulnerable populations: adults unable to consent, individuals too young to consent, prisoners, and pregnant women.
  Interventions: Combination Product: Flourish Vaginal Care System
- Study Group: 6 month study: Premenopausal women between 18 and 52 who have been diagnosed with BV at least once within the past year will be invited to enroll. They will be followed longitudinally for six months. As this is an observational study, there is no control group.
  Exclusions: pregnant women, those with allergies/sensitivities to product ingredients or to Diflucan or metronidazole, anyone who is immunocompromised, anyone with known vaginal infection other than BV or yeast, those who may be mentally/emotionally triggered by VSQ questions. We will exclude vulnerable populations: adults unable to consent, individuals too young to consent, prisoners, and pregnant women.
  Interventions: Combination Product: Flourish Vaginal Care System

INTERVENTIONS:
Combination Product: Flourish Vaginal Care System — This is not technically an intervention. All women who enroll in the study will be those who have opted to use the Flourish Vaginal Care System. This system is comprised of a vaginal wash (Balance), an intravaginal moisturizing gel (Restore), and a vaginal probiotic supplement (BiopHresh). Balance will be used daily. Restore will be used every other day. BiopHresh will be used twice a week with Restore. All products will be started after the first visit and continue throughout the 6-month study.

SUMMARY:
Background

Bacterial Vaginosis is the most common vaginal infection in women in their reproductive years and a difficult one to treat. In the United States, the National Health and Nutrition Examination Survey (NHANES), estimated the prevalence of BV was 29 percent in the general population of women aged 14 to 49 years and 50 percent in African-American women. It is characterized by a shift in vaginal flora from an acidic environment due to acid producing lactobacilli to a mixture of anaerobic and facultative microorganisms. BV causes symptoms of vaginal odor, itching, discharge and irritation and can greatly impact a woman's health, quality of life, sexual relations, self-image and well-being. BV has also been associated with an increased risk of preterm labor, STD acquisition and vaginal cuff cellulitis after hysterectomy6. After treatment with antibiotics, recurrences are common. About 15-30% will have recurrence in 3 months7.

Normal vaginal flora is lactobacilli dominant. Lactobacilli maintain vaginal pH in the acidic range and keep the growth of BV associated bacteria at low levels. Lactobacilli also produce proteins with bactericidal activity which help to maintain their dominance. Anything that alters the vaginal flora and changes the pH to a more basic environment may increase the risk of BV.

Currently, there are many sexual lubricants and vaginal moisturizers available on the market. It has recently been shown that many of these are hyperosmolar and it is thought that hyperosmolar lubricants can be damaging to the epithelium and may alter the pH of the vagina. It is postulated that lubricants and moisturizers may predispose to BV by altering the pH of the vagina.

The Flourish Vaginal Care System, by Good Clean Love, includes the following three products:

Restore, a 510K-cleared moisturizing personal lubricant that has been on the market for 3 years. It is available without a prescription. It is formulated to bio-match the vaginal secretions of women with L. crispatus-dominated microbiota. Restore has a pH of 3.7 with racemic 1% lactic acid, and is iso-osmolar with serum. It is, therefore, much less likely to alter the acid base balance of the vagina, and therefore less likely to predispose to BV.

BiopHresh Vaginal Probiotic Suppository, a Bio Matched probiotic homeopathic formulation which provides a clinically-tested combination of lactobacilli including L. crispatus and other strains found in the most stable vaginal microbiome. Research has shown as many as 30% of women do not naturally produce these critical strains of lactobacilli.

Balance Moisturizing Personal Wash is a gentle, pH-balancing cleanser with soothing botanical extracts, formulated with more than 60% premium aloe. It is made without toxic saponifiers found in most bar soaps and OTC cleansers, which tend to disrupt the cell to cell adhesion barrier8.

The aim of this study is to determine if Flourish Vaginal Care System aids in re-establishing and maintaining a healthy vaginal microbiome by restoring the vaginal pH in to the acidic range. The healthiest vaginal environments are characterized by optimal acidic vaginal pH levels, the presence of specific strains of lactobacilli. The secondary aim is to determine if the continued use of Flourish will prevent recurrence of BV over a 6 month period. The third aim is to determine what the vaginal microbiome community state type is after 6 months of Flourish use.

This study is designed to be a pilot/feasibility study. The study will compare the subjects to a historical recurrence risk7. It will also assess the ability of subjects to comply with the protocol.

DETAILED DESCRIPTION:
Methods:

Over a 2 year period, women in one academic OB/GYN clinic, who are patients of the PI and sub-investigator, with a history of at least one prior episode of BV in the past year, (confirmed via medical records) who currently have BV diagnosed via wet mount and vaginal pH, will be approached during a clinical visit regarding their desire to participate in the trial. If the subject chooses to participate after a thorough discussion of the risks and benefits, she will sign the informed consent and be enrolled in the trial. Subjects will be screened as per the providers' discretion for GC/ CH and trichomonas if it seems indicated per sexual history and/ or has not been screened in the last 3 months. A total of 40 patients will be enrolled; 20 in a shorter (12-week) preliminary study without microbiome analysis, and 20 in a longer (6-month) study including microbiome analysis.

Once enrolled, each subject will be assigned a study number by the research nurse and receive a packet of study materials from a study physician/clinician or the research nurse as well as a "Guide to Completing the BV Trial." This is a booklet containing detailed instructions for each day of the study as well as a diary in which participants will record daily symptoms. Demographic and past medical history information will also be collected at this visit.

On the first day of enrollment, subjects will be screened for BV using the Affirm VPIII test, the wet mount, vaginal pH and Nugent scoring. The Affirm test, wet mount, and vaginal pH will be done in the office, the Nugent scoring will be done by Dr. Vonetta Edwards. Subjects will also complete the vulvovaginal symptoms questionnaire (VSQ). If subjects present with either BV or yeast infection, they will be treated with standard of care. After the initial visit, all subjects will begin to use Balance every day, Restore every other day, and BiopHresh every third day until the completion of the study.

Subjects will return every 6 weeks for the remainder of the study to assess AE/SAE and test for BV the same as at the screening visit. These visits and all other study related visits will be with either the PI or sub-investigator. If the participant is found to have BV at one of these visits they will be treated using standard of care and continue using the system as directed. For subjects in the shorter study, subjects will be screened for BV/yeast, vaginal pH, and Nugent scoring every 6 weeks. For those in the longer study, at 3 months and 6 months, the subject will be rescreened for BV using the Affirm VPIII test, vaginal pH and Nugent scoring, and will complete the VSQ. At the 6 month visit, they will repeat all the same procedures and also have a vaginal swab done for analysis by the Juno Vaginal Microbiome Test. They will also be interviewed to obtain clinical experiences during the trial and will turn in a journal of daily product use and symptoms completed throughout the study. This will be obtained a member of the research team.

Monitoring of AE / SAE

The PI or sub-investigator will monitor AEs and SAEs. Sexual Health and Wellness Institute, Sponsor of the study, will not interact directly with participants but will have a staff member in the role of "Physician Liaison" available to assist physicians/clinicians at all times for the duration of the study. To maintain confidentiality, the Physician Liaison is the only Sponsor staff that will have access to patient information including patient names and patient physician names and contact information.

Study Oversight

The study may be prematurely terminated if it is determined that an abnormal number of participants experience SAEs directly associated with study materials, as verified and reported by their physician/clinician. Study Sponsor (Sexual Health and Wellness Institute) will be responsible for making this determination.

Data Management

When all participants have completed the study with the participating clinicians, participants' diaries and results of swab tests will be collected from participating clinicians, and clinical experiences during the trial will be obtained by short in person interviews by a member of the research team. Data from the participants' diaries and data obtained from interview will be analyzed.

ELIGIBILITY:
Inclusion:

Cis women aged 18-52 History of at least one prior episode of BV in the past year

Exclusion:

Pregnant Lactating Postmenopausal Immunosuppressed Known allergies to aloe vera or to other components of Restore, Balance or BiopHresh Known allergy or intolerability to po Diflucan or metronidazole Known vaginal infection that is not yeast or BV Mental/emotional triggering by sensitive questions or procedures.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Over a 2 year period, women in one academic OB/GYN clinic, who are patients of the PI and sub-investigator, with a history of at least one prior episode of BV in the past year, (confirmed via medical records) will be approached during a clinical visit regarding their desire to participate in the trial. If the subject chooses to participate after a thorough discussion of the risks and benefits, she will sign the informed consent and be enrolled in the trial. Subjects will be screened as per the providers' discretion for gonorrhea, chlamydia, and trichomonas if it seems indicated per sexual history and/ or has not been screened in the last 3 months. A total of 20 patients will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Vaginal pH Levels | 6 months
  The first aim of this study is to determine if Flourish Vaginal Care System is able to reduce the vaginal pH to a health level (pH 3.5-4.2) in order to support a healthier vaginal microbiome.
BV recurrence (assessed using Affirm VPIII test, BD Diagnostics) | 6 months
  The secondary aim is to determine if the continued use of Flourish will prevent recurrence of BV over a 6 month period. Subjects will be tested every 3 months, or more frequently if symptoms of BV or yeast infection develop.
Vaginal microbiome (assessed using the Juno Vaginal Microbiome Test, a next-generation sequencing technology) | 6 months
  This aim is to determine what the composition of the vaginal microbiome is after six months of using the Flourish Vaginal Care System in women who had recurrent BV. This is a one-time sample collection and analysis at the end of the study.

SECONDARY OUTCOMES:
Yeast infections (assessed using the Affirm VPIII test) | 6 months
  A secondary aim is to determine frequency of yeast infections while using the Flourish Vaginal Care System. Subjects will be tested every 3 months, or more frequently if symptoms of BV or yeast infection develop.
Protocol compliance via qualitative analysis of daily journal entries. | 6 months
  A secondary aim is to determine how well study subjects are able to adhere to the study protocol. This is a descriptive analysis to determine how often women follow protocol as described, and what kinds/magnitude of deviations occur.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Strgar, Study Director — Sexual Health & Wellness Institute
Locations (1):
- Concord Hospital, Concord, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nasioudis D, Linhares IM, Ledger WJ, Witkin SS. Bacterial vaginosis: a critical analysis of current knowledge. BJOG. 2017 Jan;124(1):61-69. doi: 10.1111/1471-0528.14209. Epub 2016 Jul 11. PMID 27396541
- [Background] Allsworth JE, Peipert JF. Prevalence of bacterial vaginosis: 2001-2004 National Health and Nutrition Examination Survey data. Obstet Gynecol. 2007 Jan;109(1):114-20. doi: 10.1097/01.AOG.0000247627.84791.91. PMID 17197596
- [Background] Ruiz FO, Pascual L, Giordano W, Barberis L. Bacteriocins and other bioactive substances of probiotic lactobacilli as biological weapons against Neisseria gonorrhoeae. Pathog Dis. 2015 Apr;73(3):ftv013. doi: 10.1093/femspd/ftv013. Epub 2015 Feb 11. PMID 25673666
- [Background] Edwards D, Panay N. Treating vulvovaginal atrophy/genitourinary syndrome of menopause: how important is vaginal lubricant and moisturizer composition? Climacteric. 2016 Apr;19(2):151-61. doi: 10.3109/13697137.2015.1124259. Epub 2015 Dec 26. PMID 26707589
- [Background] van de Wijgert JHHM, Jespers V. The global health impact of vaginal dysbiosis. Res Microbiol. 2017 Nov-Dec;168(9-10):859-864. doi: 10.1016/j.resmic.2017.02.003. Epub 2017 Mar 1. PMID 28257809
- [Background] Larsson PG. Treatment of bacterial vaginosis. Int J STD AIDS. 1992 Jul-Aug;3(4):239-47. doi: 10.1177/095646249200300402. No abstract available. PMID 1504154
- [Background] Ananthapadmanabhan KP, Moore DJ, Subramanyan K, Misra M, Meyer F. Cleansing without compromise: the impact of cleansers on the skin barrier and the technology of mild cleansing. Dermatol Ther. 2004;17 Suppl 1:16-25. doi: 10.1111/j.1396-0296.2004.04s1002.x. PMID 14728695